CLINICAL TRIAL: NCT01058083
Title: A Double-blind, Placebo-Controlled, Parallel-Group, Randomized, Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Effects of BMS-770767 in Subjects With Primary Hypercholesterolemia
Brief Title: Safety Study of BMS-770767 in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB117-004; 2009-014306-33 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — BMS-770767

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BMS-770767 (Treatment A) (Experimental)
  Interventions: Drug: BMS-770767
- BMS-770767 (Treatment B) (Experimental)
  Interventions: Drug: BMS-770767
- BMS-770767 (Treatment C) (Experimental)
  Interventions: Drug: BMS-770767
- BMS-770767 (Treatment D) (Experimental)
  Interventions: Drug: BMS-770767
- Placebo (Treatment E) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-770767 — Active, Oral, 15 mg, Daily, 28 days
  Arms: BMS-770767 (Treatment A)
Drug: BMS-770767 — Active, Oral, 50 mg, Daily, 28 days
  Arms: BMS-770767 (Treatment B)
Drug: BMS-770767 — Active, Oral, 150 mg, Daily, 28 days
  Arms: BMS-770767 (Treatment C)
Drug: BMS-770767 — Active, Oral, 50 mg BID, Daily, 28 days
  Arms: BMS-770767 (Treatment D)
Drug: Placebo — Placebo, Oral, 0 mg, daily, 28 days
  Arms: Placebo (Treatment E)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacodynamic effects on LDL cholesterol (LDL-C)

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemia
* Currently taking a stable daily dose of statin therapy
* Serum triglyceride level < 500mg/dl

Exclusion Criteria

* History of myocardial infarction, coronary angioplasty or bypass grafts, valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accidents within six months prior to entry into the study
* Congestive heart failure
* Diabetes mellitus
* Active liver disease
* Impaired renal function
* Hepatitis C, B and HIV

This list is not inclusive additional information is provided in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Lowering of LDL-C | Within 28 days following dosing

SECONDARY OUTCOMES:
Pharmacokinetics (Blood Level) of BMS-770767 | Within 28 days following dosing
Pharmacodynamic effects of BMS-770767 on Total cholesterol, HDL-C, Triglycerides, non-HDL-C, non-esterified free fatty acids, Apolipoprotein fractions, HPA axis marker and free testosterone and sex hormone binding globulin (SHBG) | Within 28 days following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (2):
  - Harrell, Robert, Little Rock, Arkansas
  - Cetero Research - San Antonio, San Antonio, Texas
- Australia (6):
  - Local Institution, Blacktown, New South Wales
  - Local Institution, Hornsby, New South Wales
  - Local Institution, Caboolture, Queensland
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Daw Park, South Australia
  - Local Institution, Nedlands, Western Australia
- Canada (6):
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Brampton, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Mirabel, Quebec
  - Local Institution, Montreal, Quebec

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx